CLINICAL TRIAL: NCT03082690
Title: Phase 1 Study of the Safety, Toxicity, Pharmacokinetics, Pharmacodynamics and Luminal Distribution of Single-dose DuoGel Through Rectal Administration
Brief Title: ImQuest (IQP) DuoGel Phase 1 Pharmacokinetic Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: ImQuest Pharmaceuticals, Inc. (Industry); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00041089; 5U19AI101961 (NIH)
Record Dates: First submitted 2017-03-05; First posted 2017-03-17 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: HIV Prevention
MeSH Terms: interventions — IQP-0528

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DuoGel (Experimental): IQP-0528 1% gel administered rectally one time
  Interventions: Drug: DuoGel

INTERVENTIONS:
Drug: DuoGel — 1% IQP-0528 in gel formulation
  Other Names: IQP-0528

SUMMARY:
The purpose of this study is describe the safety and single-dose pharmacokinetics of rectally-administered IQP (ImQuest Pharmaceuticals)-0528 (DuoGel) in plasma, rectal tissue biopsies, vaginal tissue biopsies, rectal fluid and cervicovaginal fluid as well as to assess the luminal distribution of IQP-0528 in the rectum. Sixteen healthy volunteers will receive a single rectal dose of DuoGel, followed by blood, tissue and fluid sampling over the following 72 hours.

DETAILED DESCRIPTION:
This is a phase 1 open label study of the safety, PK, and PD of single-dose 10 mL IQP-0528 through rectal administration. Pharmacokinetics (PK) will be assessed in multiple compartments: plasma, rectal tissue, vaginal tissue, rectal fluid and cervicovaginal fluid. The luminal distribution of DuoGel in the rectum will be evaluated with Single Photon Emission Computed Tomography/ X-ray Computed Tomography (SPECT/CT). Pharmacodynamics (PD) will be assessed in an ex vivo HIV explant challenge of rectal and vaginal tissue biopsies.

After completing the screening evaluation (Visit 1) and establishing participant eligibility, 16 eligible participants will be enrolled: 8 men and 8 women. A subsequent baseline visit (Visit 2) safety assessment and tissue ex vivo HIV explant challenge will be performed as baseline for comparison with later post-drug evaluation. Participants will receive a single 10 mL rectal dose of 99mTechnetium (99mTc) -radiolabelled DuoGel (Visit 3), followed by safety assessments and PK and PD sampling over three days (Visits 3, 4, and 5). Finally, a follow-up safety phone call is performed a week after all PK sampling and biopsies are collected.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older at screening
* HIV-1 negative as documented at screening
* Willing to use condoms for the duration of the study
* Willing to refrain from aspirin and non-steroidal anti-inflammatory drug (NSAID) use for one week before and after each study biopsy visit
* Available to return for all study visits
* Agrees to sexually transmitted infection (STI) reporting requirements
* Able and willing to communicate in English
* Able and willing to provide written informed consent
* Able and willing to provide adequate information for locator purposes
* Agrees not to participate in other research studies
* Willing to refrain from receptive anal intercourse and insertion of anything in the rectum for 72 hours before and after rectal biopsies.

Additional inclusion criteria for women:

* Be pre-menopausal
* Have regular menstrual cycles (unless on contraception that causes amenorrhea or irregular menses)
* Have a negative qualitative urine pregnancy test
* Per participant report, using an effective method of contraception at enrollment; hormonal method (except vaginal ring) used continuously for the past 30 days; intrauterine device (IUD [copper or hormonal] inserted at least 30 days prior to enrollment); female sterilization; abstinent from sexual activity with male partner for the past 30 days; or sexual activity with vasectomized partner; and willingness to use effective method of contraception until the completion of final scheduled study visit if enrolled.
* Willing to refrain from insertion of anything into the vagina for at least 72 hours before and 7 days after vaginal biopsies.

Exclusion Criteria:

* Current known HIV-infected partners
* Current use of anticoagulant medications associated with increased risk for bleeding following mucosal biopsy (e.g., daily high dose aspirin [>81 mg], NSAIDs, or Pradaxa®)
* Current use of cytochrome P450 3A (CYP3A) inducer(s) and/or inhibitor(s)
* Use of systemic immunomodulatory medications within 4 weeks of enrollment
* Known allergic reaction to components of the study product
* History of recurrent urticaria
* Participants whose whole body radiation exposure exceeds 5000 millirem (mRem)/year.
* Participants who are currently receiving or have been on oral PrEP or PEP in the past month
* Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study or unable to comply with the study requirements.
* Significant colorectal symptom(s) as determined by medical history or by participant self-report
* Active rectal infection, requiring treatment per current Centers for Disease Control (CDC) guidelines or symptomatic urinary tract infection (UTI). Infections requiring treatment include Chlamydia (CT), gonorrhea (GC), syphilis, active herpes simplex virus (HSV) lesions, chancroid, genital sores or ulcers, and, if clinically indicated, genital warts.
* History of STI within the last 3 months.
* Use of post-exposure (PEP) or pre-exposure (PrEP) prophylaxis within the last 6 months
* History of significant gastrointestinal bleeding
* Use of any rectally administered medications within 4 weeks of enrollment or unwillingness to refrain from use of any rectally administered medications 72 hours prior to any study dosing or biopsy visit
* Use of any rectally administered products containing nonoxynol-9 (including condoms) or investigational products within 4 weeks of enrollment

Additional exclusion criteria for women:

* Significant vaginal symptoms, genital lesions, erythema, edema or any other abnormal physical finding that, in the opinion of the investigator or designee, would contraindicate study participation.
* Active female genital tract infection, requiring treatment per current CDC guidelines or symptomatic urinary tract infection (UTI). Infections requiring treatment include Chlamydia (CT), gonorrhea (GC), syphilis, active HSV lesions, chancroid, bacterial vaginosis, vaginal candidiasis, trichomonas, genital sores or ulcers, and, if clinically indicated, genital warts.
* History of significant vaginal bleeding
* Undiagnosed irregular uterine bleeding
* Post-menopausal defined as 12 months of amenorrhea
* Per participant report, abnormalities of the female genital tract, which, in the judgment of the investigator, might increase the risk of the study to the research participant.
* Per participant report, history of cervical procedures (conization, Loop El electrosurgical Excision procedure (LEEP) procedure, cryosurgery) within the previous 6 months.
* Per participant report, use of any vaginally administered medications within 4 weeks of enrollment
* Per participant report, use of any vaginally administered products containing nonoxynol-9 (including condoms) or investigational products within 4 weeks of enrollment
* Women who are pregnant or breastfeeding
* Spermicide use within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-06-02 (Actual)

PRIMARY OUTCOMES:
To assess systemic and local safety of 10 mL of IQP-0528 following rectal administration by adverse events. | One week
  Grade 2 or above adverse events as measured by the Division of AIDS Toxicity Table
To assess rectal PK of 10 mL of IQP-0528 | 72 hours
  Maximum Concentration (Cmax)
To assess rectal PK of 10 mL of IQP-0528 | 72 hours
  Time to Maximum Concentration (Tmax)
To assess rectal PK of 10 mL of IQP-0528 | 72 hours
  Area Under the Curve (AUC)
To assess rectal PK of 10 mL of IQP-0528 | 72 hours
  Terminal elimination half-life

SECONDARY OUTCOMES:
To compare rectal PK between men and women | 72 hours
  Maximum Concentration (Cmax)
To compare rectal PK between men and women | 72 hours
  Time to Maximum Concentration (Tmax)
To compare rectal PK between men and women | 72 hours
  Area Under the Curve (AUC)
To compare rectal PK between men and women | 72 hours
  Terminal elimination half-life

CONTACTS AND LOCATIONS:
Overall Officials: Craig Hendrix, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al-Khouja A, Shieh E, Fuchs EJ, Marzinke MA, Bakshi RP, Hummert P, Ham AS, Buckheit KW, Breakey J, Weld ED, Chen H, Caffo BS, Buckheit RW, Hendrix CW. Examining the Safety, Pharmacokinetics, and Pharmacodynamics of a Rectally Administered IQP-0528 Gel for HIV Pre-Exposure Prophylaxis: A First-In-Human Study. AIDS Res Hum Retroviruses. 2021 Jun;37(6):444-452. doi: 10.1089/AID.2020.0188. Epub 2021 Jan 25. PMID 33371779